CLINICAL TRIAL: NCT04345224
Title: The Effect of Dynamic and Rigid Tape Application on the Asymmetry of the Lower Limbs in Healthy People
Brief Title: The Effect of Dynamic and Rigid Tape Application on the Asymmetry of the Lower Limbs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Paul II University in Biała Podlaska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PopeJohnPaulIIStateSchHigherE1
Record Dates: First submitted 2020-04-07; First posted 2020-04-14 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2021-03

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: The study participants will be randomly qualified (allocated via a computer program) to the tree groups: A - dynamic tape, B - rigid tape, C - sham tape
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dynamic tape (Experimental): The gluteal muscle group will be covered with a dynamic tape.
  Interventions: Other: Dynamic tape
- Rigid tape (Experimental): The gluteal muscle group will be covered with a rigid tape.
  Interventions: Other: Rigid tape
- Sham tape (Sham Comparator): The gluteal muscle group will be covered with a paper tape - a sham application.
  Interventions: Other: Sham tape

INTERVENTIONS:
Other: Dynamic tape — A kinesiology tape will be applied to the lateral hip of the affected side to facilitate the gluteus medius muscle activation while the participant is lying down. The first third of one I-strip will begin at the posterior iliac crest without tension to provide an anchor that will not cross the target tissue. The participant will actively flex the adducted hip to allow for the application of the middle third of the tape with approximately 50 percent tension (able to visualize the wave pattern in the tape). Subsequently, with the leg in the original position, the remainder of the tape will be applied without tension, ending approximately at the greater trochanter. Afterward, the second I-strip will be applied in the same manner starting at the anterior iliac crest.
  Arms: Dynamic tape
Other: Rigid tape — The rigid tape will be applied in a standing position. The first tape will be applied from the greater trochanter to the anterior iliac crest. The second from the greater trochanter to the posterior iliac crest. Both tapes are applied with the muscle mass lifted towards the iliac crest.
  Arms: Rigid tape
Other: Sham tape — The control group (sham tape application) will receive a single strip of a Kinesio tape across the lateral affected hip without tension in the tape or muscle stretch.
  Arms: Sham tape

SUMMARY:
This is a prospective randomized three brachial, single-blinded, placebo-controlled trial, which aims at assessing the impact of the gluteal muscle taping with a dynamic tape and a non-elastic tape on the activation of the gluteal muscles and the distribution of the lower limb load in healthy people.

The study participants will be randomly classified into the following groups: A - dynamic kinesiology taping, B - rigid tape, C - placebo group (sham). Patients will be evaluated three times - before applying the tapes, 30 minutes after applying the tapes and 48 hours after applying the tapes.

DETAILED DESCRIPTION:
The gluteus maximus is the largest and strongest muscle in the human body. Its function is primarily to extend the hip joint. The back fibers of the gluteus medius and gluteus minimus muscles provide the additional help. These muscles also perform the functions of abductors and external rotators of the hip joint.

The incorrect strength and activation time of the muscles stabilizing the hip joint result in the disturbed load distribution of the lower limbs. This may cause the overloading of the bone and muscle structures. Disorders of the functions of the external hip rotators and abductors may lead to such health problems as: patellofemoral conflict, ilio-tibial band syndrome or non-specific pains of the hip, knee, sacroiliac and lumbar spine. Neurological diseases, such as stroke, causing paresis of the limbs, accompanied by a decrease or increase in muscle tone and disturbed load distribution, are also an obstacle to gait re-education and limit the efficiency of everyday activities.

Dynamic tapes were created by Kenso Kase MD in Japan. Their characteristic feature is extensibility reaching 130-140 percent. The tape is based on sensory effects on fascia mechanoreceptors. Depending on the slicing technique used, the following effects can be achieved: the activation or reduction of muscle tone, the reduction of pain and an increased flow of tissue fluids.

The concept of using a rigid tape was created and developed by Jenny McConnell. A characteristic feature of a rigid tape is the lack of stretchability, thanks to which mechanical stabilization of a specific section of the body can be achieved. The effects of using a rigid tape include: the reduction of pain, the activation or reduction of muscle tone, and the correction of joint components.

For many years, research has been conducted into the effects of using a dynamic tape and a rigid tape on the muscle functions. In many cases, reports from various authors are contradictory. There is also a lack of publications assessing the effect of a tape on the buttock muscle activation and the associated lower limb load distribution. There is therefore a need for further research.

The aim of the project is to assess the impact of gluteal muscle taping with a dynamic tape and a rigid tape on the distribution of lower limb load in healthy people. The confirmation of research hypotheses will allow for the introduction of a new therapy tool in neurological patients (e.g. after stroke), but also healthy people, to prevent a lower limb and spine structures overloading.

ELIGIBILITY:
Inclusion Criteria:

* not using non-steroidal anti-inflammatory drugs (NSAIDs) for at least one week prior to testing,
* age - 19-24 years old

Exclusion Criteria:

* spine, hip, knee or ankle surgery,
* spine, hip, knee or ankle injuries within 6 months before the start of the examination,
* neurological and otolaryngological diseases, which may result in imbalances.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Tests on the dynamographic platform | Before applying the tape and after 2 days
  Assessment of:
  * the lower extremity load when standing with eyes open,
  * the lower extremity load when standing with eyes closed,
  * the lower limb load when walking in place,
  * the lower limbs loading when sitting and getting up from a chair. The symmetry index (Ws) will be calculated from the result of each test.The symmetry index calculated as the quotient of the load results of a more heavily loaded limb to a less loaded limb. The correct value of the indicator is taken from 1.0 to 1.15.
Muscle activation test using NaroxonUltium (EMG) - Maximum Voluntary Isometric Contraction (MVIC) | Before applying the tape
  The gluteus medius muscle MVIC will be performed while lying on one's side, with the hip in a neutral rotation and slightly extended and then actively abducted to end range as resistance will be applied just above the ankle.The maximal hip abductor strength will be tested 3 times per leg for each participant.The maximal strength will be defined as the peak force recorded by the digital force gauge.
Muscle activation test using NaroxonUltium (EMG) - Unilateral bridge | Before applying the tape and after 2 days
  Participant is in a supine position with the bilateral knees bent at 90 degrees.Participant lifts the leg and extends it at the knee,then lifts the bilateral hips to the neutral hip position with the right leg only.
  The results of the test (the peak force) will be calculated and presented as percentage MVIC.
Muscle activation test using NaroxonUltium (EMG) - Side-lying hip abduction | Before applying the tape and after 2 days
  Participant is lying on their side with the bottom leg bent to keep the body form rotating.The top leg is abducted approximately at 25 degrees, held for 2-3 seconds and adducted to the starting position. The results of the test (the peak force) will be calculated and presented as percentage MVIC.

CONTACTS AND LOCATIONS:
Overall Officials: Krystyna Gawlik, Ph.D, Study Chair — Pope John Paul II State School of Higher Education in Biala Podlaska
Locations (1):
- Pope John Paul II State School Of Higher Education in Biała Podlaska, Biała Podlaska, Poland

IPD SHARING:
Plan to Share IPD: No